CLINICAL TRIAL: NCT04275557
Title: Using Radiogenomics to Noninvasively Predict the Malignant Potential of Intraductal Papillary Mucinous Neoplasms (IPMNs) of the Pancreas and Uncover Hidden Biology
Brief Title: Using Radiogenomics to Predict Malignant Potential of Intraductal Papillary Mucinous Neoplasms of the Pancreas
Status: Recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Florida (Other); University of Miami (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-20105; 1R37CA229810-01A1 (NIH)
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer; Pancreatic Cyst
Keywords: Pancreatic Lesions
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Cyst | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole Blood, Plasma, Serum, Tumor tissue from biopsy or surgery, Muscle and fat tissue from surgery, cyst fluid, cytology supernatant, peripheral blood monocular cells (PMBCs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Cohort: Retrospective chart review of pathologically-confirmed Intraductal Papillary Mucinous Neoplasm (IPMN) cases
- Prospective Cohort: Blood, tumor tissue samples and data will be collected.
  Interventions: Other: Blood Sample collection; Other: Tissue sample collection; Other: Data collection

INTERVENTIONS:
Other: Blood Sample collection — Participants will be asked to donate blood at baseline (+/- 30 days of diagnosis date), 4-6 weeks post-surgery, if applicable, and at the time of follow-up (approximately 1 year and approximately 2 years after baseline).
  Groups: Prospective Cohort
Other: Tissue sample collection — At the time of tissue biopsy and surgical resection (if applicable), pancreatic tumor tissue, muscle, fat, tissue from site of metastasis, and cyst fluid (if applicable) will be collected.
  Groups: Prospective Cohort
Other: Data collection — Participants will be asked to complete questionnaires at baseline and at 1 year and 2 year follow-ups.
  Groups: Prospective Cohort

SUMMARY:
The Florida Pancreas Collaborative wants to partner with individuals who are known to have, or are suspected to have a pancreatic lesion, tumor, cyst, mass, cancer, or pancreatitis and are undergoing diagnosis and treatment at a participating institution. The goals of this project are to build a large database of information obtained from blood, tissue, medical images, surveys and information from routine care to develop noninvasive diagnostic approaches that could be used as decision-making tools to effectively personalize clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who present to the GI clinic, surgery, or endoscopy at Moffitt, Florida Research Institute (FRI), or UM with a clinical suspicion for (or diagnosis of) a pancreatic lesion, cyst, mass, cancer, or pancreatitis based on symptoms, imaging, or blood-work and has not had any treatment involving their pancreas.
* Able to understand and voluntarily sign the informed consent.
* Willing to complete study questionnaire(s) and donate medical images and/or biological specimens (including blood, cystic fluid, and/or tissue) obtained at the time of standard of care procedures (biopsy, surgery, and venipuncture) after signing the informed consent document

Exclusion Criteria:

* No suspicion or diagnosis of a pancreatic lesion, cyst, mass, cancer, or pancreatitis.
* Has a diagnosis of a pancreatic lesion, cyst, mass, cancer, or pancreatitis and has already undergone treatment involving the pancreas (which may involve surgery, chemo- or immuno-therapy, and/or radiation).
* Unable to provide informed consent.
* Unwilling to complete study questionnaire(s) and/or donate biological specimens or images.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the GI clinic, surgery, or endoscopy at Moffitt Cancer Center, University of Florida - Gainesville, or the University of Miami - Jackson Memorial Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1174 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Predictive value of CT Radiomic features vs conventional radiologic features | Up to 2 years
  Preoperative CT images will be evaluated for a retrospective cohort of at least 254 pathologically-confirmed IPMN cases (approximately 190 malignant characterized by high-grade dysplasia or invasion and approximately 64 benign characterized by low- or moderate-grade dysplasia). 3D-radiomic features will be extracted with the new Quantitative Imaging Decision Support (QIDS)™ platform (Healthmyne, Inc.) and associations will be evaluated with pathology.
Development of Clinical Decision Making Models for Predicting IPMN Pathology | Up to 2 years
  Investigators will develop the first prototype preoperative 'omics'-based nomograms to predict IPMN pathology by integrating radiomic features, the MGC, and other covariates. Emphasis will be placed on developing nomograms for individuals whose IPMNs appear to have 'worrisome' radiologic features which are very challenging to manage.
Radiogenomic Analyses | Up to 2 years
  Investigators will conduct the first radiogenomic analyses of IPMNs by evaluating the relationship between radiomic features and tissue and circulating levels of candidate biomarkers.

SECONDARY OUTCOMES:
Overall Survival | Up to 4 years
  Overall survival is defined as time from surgery to death from any cause.
Progression Free Survival | Up to 4 years
  Progression free survival is defined as time from surgery to either pancreatic cancer recurrence or death.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Permuth, PhD, Principal Investigator — Moffitt Cancer Center
Locations (3):
- United States (3):
  - Florida Research Institute (FRI), Lakewood Rch, Florida
  - Sylvester Comprehensive Cancer Center & Jackson Memorial Hospital, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Moffitt Cancer Center website — http://www.moffitt.org